CLINICAL TRIAL: NCT02747706
Title: Peer Mentor Training to Reduce Hospitalizations for Children With Asthma
Brief Title: Childhood Asthma Mentoring Program for Parents
Acronym: CAMPP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: InquisitHealth, Inc. (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Montefiore Medical Center (Other); University of North Carolina, Chapel Hill (Other); Washington University School of Medicine (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Ashwin Patel, Chief Medical Officer, InquisitHealth, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Asthma23; 4R44HD081830 (NIH)
Record Dates: First submitted 2016-04-18; First posted 2016-04-22 (Estimated); Last update posted 2016-04-22 (Estimated); Status verified 2016-04

CONDITIONS: Asthma
Keywords: peer mentor; health coach; parent support; parent mentor
MeSH Terms: conditions — Asthma

ARMS (2):
- Parent Mentoring (Experimental): 1-on-1, phone, SMS/text, and smartphone-based parent-to-parent mentoring.
  Interventions: Behavioral: Parent-to-parent mentoring
- Usual Care (No Intervention): No intervention through study.

INTERVENTIONS:
Behavioral: Parent-to-parent mentoring — phone, SMS/text, and smartphone-based support
  Arms: Parent Mentoring

SUMMARY:
There are 7.1 million children with asthma. Asthma is the cause of 10.5 million missed days of school, 7.5 million outpatient visits, 640,000 ED visits, and 157,000 hospitalization visits in 2008. Recent work has demonstrated that trained peer mentors (individuals from the community) can be effective in reducing hospitalizations for asthmatic children.

This study will evaluate the efficacy of technology-driven parent-to-parent mentoring to reduce asthma-related pediatric hospitalizations and emergency department visits.

ELIGIBILITY:
Inclusion Criteria:

* Parent of child with persistent asthma, prescription of controller medications, and at least one asthma exacerbation in the past year

Exclusion Criteria:

* Parent has no access to smartphone

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 240 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-09 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Number of hospital admissions | 1-year
Number of emergency department visits | 1-year

CONTACTS AND LOCATIONS:
Overall Officials: Ashwin Patel, MD PhD, Principal Investigator — Chief Medical Officer
Locations (1):
- InquisitHealth, River Edge, New Jersey, United States